CLINICAL TRIAL: NCT04786093
Title: Randomized Phase II Study of Durvalumab (MEDI 4736) and Stereotactic Radiotherapy for Advanced Non-Small Cell Lung Cancer
Brief Title: Durvalumab and Stereotactic Radiotherapy for Advanced NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Shahed Badiyan, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0171
Record Dates: First submitted 2021-02-28; First posted 2021-03-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Immunotherapy; Durvalumab; Radiation therapy; Radiotherapy; Stereotactic body radiation therapy; Stereotactic ablative radiotherapy; SBRT; SABR; PULSAR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; durvalumab

STUDY DESIGN:
Intervention Model Description: We hypothesize that Durvalumab and stereotactic radiotherapy, in the form of PULSAR and SAbR, and durvalumab will confer a 60% increase in improvement in quality of life over the historical control rate of 33%, for an absolute improvement of 27%. Using a two-sided exact binomial test with a two-sided significance level of 0.1 and 80% power, we estimate that we will need to enroll 23 patients per arm do detect a difference. Accounting for 10% attrition, we will plan to enroll 52 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stereotactic Ablative Radiotherapy (SAbR) Arm plus Durvalumab arm (Active Comparator): SAbR with each radiation treatment fraction delivered every other day
  Interventions: Radiation: Stereotactic radiation therapy; Drug: Durvalumab
- Personalized Ultra-fractionated Stereotactic Radiotherapy (PULSAR) plus Durvalumab arm (Experimental): PULSAR with each radiation treatment fraction delivered every 4 weeks
  Interventions: Radiation: Stereotactic radiation therapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Stereotactic radiation therapy — Radiation therapy will be delivered using standard SAbR treatment schedule or every 4 weeks on the PULSAR schedule to achieve optimal local control of metastatic cancer and augment the effects of durvalumab.
Drug: Durvalumab — Durvalumab (initially developed as MEDI4736) is a human monoclonal antibody of the immunoglobulin (Ig) G1 kappa subclass that inhibits binding of PD-L1 (B7-H1, CD274) to PD-1 (CD279) and CD80 (B7-1). MEDI4736 is composed of 2 identical heavy chains and 2 identical light chains, with an overall molecular weight of approximately 149 kDa. MEDI4736 contains a triple mutation in the constant domain of the Ig G1 heavy chain that reduces binding to complement protein C1q and the fragment crystallizable gamma receptors involved in triggering effector function.

SUMMARY:
This is a randomized Phase II study which is designed to determine the impact of stereotactic radiotherapy and durvalumab on quality-of-life and oncologic outcomes in patients with advanced non-small cell lung cancer. Durvalumab (Imfinzi) and stereotactic radiotherapy, with each fraction of radiotherapy is given every other day on a standard stereotactic ablative radiotherapy (SAbR) schedule or every four weeks on the personalized ultra-fractionated stereotactic adaptive radiotherapy (PULSAR) schedule. Subjects will be followed for a period of 2 years after completion of treatment or until death, whichever occurs first. Specifically, subjects will be followed at 1, 3, 6, 9, 12, 15, 18, 21, and 24 months following treatment. After the 2 year follow up, the patient can continue routine follow up with their physicians, per standard of care. Subjects removed from therapy for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy-proven metastatic non-small cell lung cancer and eligible for receipt of immunotherapy, based on standard of care
2. Patients can present with either de novo metastatic disease or recurrent disease
3. Patients must have at least one (1) symptomatic or progressive metastatic sites with no more than 10 metastatic sites, based on standard imaging studies
4. Patients cannot have received any prior radiation therapy or surgery to the intended radiation treatment area (index lesion)
5. Patients with brain metastases may be enrolled if all lesions are treated with radiation therapy or surgery prior to start of protocol therapy
6. Metastases in major lower extremity weight-bearing bones or spine should undergo surgical stabilization if indicated
7. Age greater than or equal to 18 years.
8. Both men and women and members of all races and ethnic groups will be included
9. Eastern Cooperative Oncology Group Performance status 0 to 2 (Appendix A)
10. Adequate normal organ and bone marrow function as defined by:

    * Haemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1.0 × 109 /L
    * Platelet count ≥75 × 109/L
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * AST (SGOT)/ALT (SGPT) ≤2.5X institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5X ULN
    * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

      1. Males:

         * Creatinine CL (mL/min) = (Weight (kg) x (140 - Age)) ÷ (72 x serum creatinine (mg/dL))
      2. Females:

         * Creatinine CL (mL/min) = ((Weight (kg) x (140 - Age)) ÷ (72 x serum creatinine (mg/dL))) x 0.85
11. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

    Medically accepted forms of birth control include male condoms plus spermicide, diaphragm, cervical cap, the placement of a Copper T intrauterine device (IUD), birth control pills, Levonorgesterel-releasing intrauterine system (IUS), hormone implants or injections, or combined pill, minipill patch, or a partner who has undergone a vasectomy (surgical sterility).
    * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

      * Has not undergone a hysterectomy or bilateral oophorectomy; or
      * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
12. Life expectancy greater than six (6) months
13. Body weight greater than 30 kg
14. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
15. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
2. Administration of two or more lines of systemic therapy for the diagnosis of metastatic non-small cell lung cancer

   * Prior receipt of systemic therapy for the management of high-risk early stage or locally advanced non-small cell lung cancer, prior to the development of metastatic disease, would not count towards the number of receipt of systemic therapy
3. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
4. Patients with untreated brain metastases
5. Patients with progressive metastatic disease involving the skin or subcutaneous tissues, esophagus, stomach, intestines, or mesenteric lymph nodes that are felt to be too high risk to treat with radiation therapy to protocol dose.
6. Patients cannot have pathologic fracture at the evaluated site
7. Patients cannot have untreated spinal cord compression
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab or other agents used in study
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
10. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
11. Male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
12. Participation in another clinical study with an investigational product during the last 3 months
13. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
14. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤7 days prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator
15. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

    * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
16. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
17. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of immunotherapy. Note: Local surgery of isolated lesions for palliative intent is acceptable
18. History of allogenic organ transplantation
19. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of immunotherapy and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo malignant without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
20. History of leptomeningeal carcinomatosis
21. History of active primary immunodeficiency
22. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
23. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
24. Receipt of live attenuated vaccine within 30 days prior to the first dose of immunotherapy. Other forms of vaccines, such as mRNA, recombinant protein, and non-replicating vector-based vaccines, are permitted. Note: Patients, if enrolled, should not receive live vaccine whilst receiving immunotherapy and up to 30 days after the last dose of immunotherapy
25. Receipt of any medications listed below:

    * Patients on this study should not be on any targeted systemic therapies such as those directed at EGFR mutations, ALK or ROS1 gene rearrangements, BRAF V600E mutation, or NTRK gene fusions. Other anti-cancer treatments are also not allowed on the study and are listed below. Supportive medications may be given at any point during treatment at the discretion of the treating physician, such as anti-emetics, pain medications, anti-diarrheals, nutritional supplementations, and anti-depressants. Anti-oxidant medications in excess of daily recommended values are not allowed.

      * Any investigational anticancer therapy other than those under investigation in this study should not be given concomitantly whilst the patient is on study treatment.
      * mAbs against CTLA-4, PD-1, or PD-L1 other than those under investigation in this study should not be given concomitantly whilst the patient is on study treatment.
      * Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment other than those under investigation in this study should not be given concomitantly whilst the patient is on study treatment. (Concurrent use of hormones for non-cancer-related conditions [e.g., insulin for diabetes and hormone replacement therapy] is acceptable. Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable [e.g., by local surgery or radiotherapy])
      * Immunosuppressive medications including, but not limited to, systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent, methotrexate, azathioprine, and tumor necrosis factor-α blockers.

        * Immunosuppressive medications should not be given concomitantly, or used for premedication prior to the IO infusions. The following are allowed exceptions:

          1. Use of immunosuppressive medications for the management of IP-related AEs,
          2. Use in patients with contrast allergies.
          3. In addition, use of inhaled, topical, and intranasal corticosteroids is permitted.
        * A temporary period of steroids will be allowed if clinically indicated and considered to be essential for the management of non-immunotherapy related events experienced by the patient (e.g., chronic obstructive pulmonary disease, radiation, nausea, etc.).
      * EGFR tyrosine kinase inhibitors (TKI) should not be given concomitantly, and should be used with caution in the 90 days post last dose of durvalumab. Increased incidences of pneumonitis (with third generation EGFR TKIs) and increased incidence of transaminase increases (with 1st generation EGFR TKIs) has been reported when durvalumab has been given concomitantly.
      * Live attenuated vaccines should not be given through 30 days after the last dose of IP (including SoC)
      * Herbal and natural remedies which may have immune-modulating effects should not be given concomitantly unless agreed by the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scores | 2 years post-treatment
  To assess the impact of durvalumab and stereotactic radiotherapy, in the form of stereotactic ablative radiotherapy (SAbR) or personalized ultra-fractionated stereotactic adaptive radiotherapy (PULSAR), on improving QoL (quality of life) in patients with metastatic non-small cell lung cancer using the European organization for Research and treatment of cancer questionnaire (EORTC-QLQ30). The score range is 0-100. Higher the score, the better the results.

SECONDARY OUTCOMES:
Local control (LC) | 1 year post-treatment
  To determine the effect of PULSAR or SAbR plus durvalumab on local control. Local control is defined as the percentage of tumors without tumor failure within the irradiated field, as defined as growth on diagnostic imaging studies or evidence of viable cancer cells. Probability will be assessed using the Kaplan-Meier method.
Out-of-field control | 1 year post-treatment
  To assess the effect of PULSAR or SAbR plus durvalumab on out-of-field control (termed abscopal response). Out-of-field control is defined as the percentage of tumors without tumor failure outside of the irradiated field, as defined as growth on diagnostic imaging studies or evidence of viable cancer cells. Probability will be assessed using the Kaplan-Meier method.
Progression free survival (PFS) | 2 years post-treatment
  To determine the effect of PULSAR or SAbR plus durvalumab on progression-free survival. Progression-free survival (PFS) is defined as the time from random assignment to disease progression or death from any cause. Probability will be assessed using the Kaplan-Meier method.
Overall Survival | 2 years post-treatment
  To determine the effect of PULSAR or SAbR plus durvalumab on overall survival. Overall survival (OS) is defined as the defined as the time between the date of randomization and the date of death due to any cause. Probability will be assessed using the Kaplan-Meier method.
overall response rate (ORR) | 12 weeks from randomization
  To determine the effect of PULSAR or SAbR plus durvalumab on overall response rate at 12 weeks. Overall response rate is defined as complete response and partial response at 12 weeks (about 3 months) from randomization.
Instances of Toxicity | 2 years post-treatment
  To determine the effect of PULSAR or SAbR plus durvalumab on toxicity. Toxicity will be assessed using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Only adverse events assessed to be definitely, probably, or possibly related to protocol treatment will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Shahed Badiyan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No